CLINICAL TRIAL: NCT00234260
Title: Family Blood Pressure Program - GENOA (Genetic Epidemiology Network of Atherosclerosis)
Status: Terminated | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: U01HL075572 (NIH)
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Last update posted 2008-07-16 (Estimated); Status verified 2005-10

CONDITIONS: Arteriosclerosis; Hypertension; Heart Diseases
Keywords: Genetics
MeSH Terms: conditions — Arteriosclerosis; Hypertension; Heart Diseases

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
GENOA, the Genetic Epidemiology Network of Arteriopathy, consists of a network of three field centers and biochemical and genetic core labs to study the common polymorphic genetic variations to determine individual differences in blood pressure and essential hypertension in 1,500 sibling pairs in three racial groups. Linkage analyses are performed using an extensive array of candidate genes and anonymous markers throughout the genome.

DETAILED DESCRIPTION:
Each collaborating investigator is responsible for an essential element of the network: Eric Boerwinkle for genotyping and linkage analyses, Robert Ferrell for genotyping, Craig Hanis for recruiting Mexican-Americans, Richard Hutchinson for recruiting African-Americans, Sharon Kardia for cladistic and prediction analyses and data management, and Stephen Turner for recruiting Non-Hispanic whites and measuring physiologic variables. Between 1995 and 2000, the network carried out five specific aims to localize and characterize the genetic determinants of high blood pressure. Aim 1 used robust sibling pair linkage methods in 500 hypertensive sibling pairs in each racial group (a total of 1,500 sibling pairs) to localize genes influencing interindividual differences in the occurrence of essential hypertension. Aims 2 and 3 took advantage of previously collected blood pressure and intermediate predictor trait data from 1,488 normotensive sibling pairs from the Rochester Family Heart Study to localize genes contributing to essential hypertension. The linkage analyses (Aims 1-3) used both an extensive array of candidate genes and a large number of anonymous markers throughout the genome. Aim 4 used multiple diallelic sequence polymorphisms and cladistic analyses within a linked gene to identify haplotypes for further DNA sequencing in order to identify candidate functional DNA sequence variation contributing to interindividual differences in BP levels and essential hypertension status. Aim 5 evaluated the ability of candidate functional DNA sequence variation to predict essential hypertension status in the three racial groups.

The study was renewed in September 2000 to pursue two lines of investigation. The first is to identify and characterize genes contributing to atherosclerotic coronary heart disease using electron beam computed tomography (EBCT) to quantify coronary artery calcification as a measure of preclinical disease. Robust sibling-pair linkage methods will be used to determine whether any of the more than 375 highly polymorphic tandem repeat marker loci spanning the genome are linked to genes influencing EBCT measures of coronary artery calcification in at least 500 GENOA sibships from Rochester, Minnesota. Association analysis will be used to determine whether biallelic markers of DNA sequence variation in candidate genes identified by GENOA or others to influence blood pressure level or diagnostic category also influence EBCT measures of coronary artery calcification in at least 500 GENOA participants from Rochester, Minnesota. The second line of investigation extends analytical methods (linkage disequilibrium regression and combinatorial partitioning) to more finely localize positional candidate genes and loci, and to identify gene-gene and gene-environment interaction effects influencing the measured Family Blood Pressure Program and GENOA phenotypes.

ELIGIBILITY:
Inclusion Criteria:

Jackson Mississippi - age 45-64, Hypertensive Rochester, Minnesota - <60, Hypertensive Starr County, Texas - <60, type II diabetes mellitus

Exclusion Criteria:

-

Max Age: 64 Years | Sex: All
Age Groups: Child, Adult
Dates: Start 1995-04

CONTACTS AND LOCATIONS:
Overall Officials: Eric Boerwinkle, PhD, Principal Investigator — Human Genetics Center, The University of Texas at Houston Health Science Center
Locations (3):
- United States (3):
  - Rochester Field Center, Rochester, Minnesota
  - Jackson Field Center, Jackson, Mississippi
  - Starr County Field Center, Rio Grande City, Texas

REFERENCES:
- [Background] FBPP Investigators. Multi-center genetic study of hypertension: The Family Blood Pressure Program (FBPP). Hypertension. 2002 Jan;39(1):3-9. doi: 10.1161/hy1201.100415. PMID 11799070
- [Result] An P, Freedman BI, Hanis CL, Chen YD, Weder AB, Schork NJ, Boerwinkle E, Province MA, Hsiung CA, Wu X, Quertermous T, Rao DC. Genome-wide linkage scans for fasting glucose, insulin, and insulin resistance in the National Heart, Lung, and Blood Institute Family Blood Pressure Program: evidence of linkages to chromosome 7q36 and 19q13 from meta-analysis. Diabetes. 2005 Mar;54(3):909-14. doi: 10.2337/diabetes.54.3.909. PMID 15734873
- [Result] Daniels PR, Kardia SL, Hanis CL, Brown CA, Hutchinson R, Boerwinkle E, Turner ST; Genetic Epidemiology Network of Arteriopathy study. Familial aggregation of hypertension treatment and control in the Genetic Epidemiology Network of Arteriopathy (GENOA) study. Am J Med. 2004 May 15;116(10):676-81. doi: 10.1016/j.amjmed.2003.12.032. PMID 15121494
- [Result] Kullo IJ, Bailey KR, Bielak LF, Sheedy PF 2nd, Klee GG, Kardia SL, Peyser PA, Boerwinkle E, Turner ST. Lack of association between lipoprotein(a) and coronary artery calcification in the Genetic Epidemiology Network of Arteriopathy (GENOA) study. Mayo Clin Proc. 2004 Oct;79(10):1258-63. doi: 10.4065/79.10.1258. PMID 15473406
- [Result] Kullo IJ, Bailey KR, Kardia SL, Mosley TH Jr, Boerwinkle E, Turner ST. Ethnic differences in peripheral arterial disease in the NHLBI Genetic Epidemiology Network of Arteriopathy (GENOA) study. Vasc Med. 2003 Nov;8(4):237-42. doi: 10.1191/1358863x03vm511oa. PMID 15125483
- [Result] Morrison AC, Cooper R, Hunt S, Lewis CE, Luke A, Mosley TH, Boerwinkle E. Genome scan for hypertension in nonobese African Americans: the National Heart, Lung, and Blood Institute Family Blood Pressure Program. Am J Hypertens. 2004 Sep;17(9):834-8. doi: 10.1016/j.amjhyper.2004.04.009. PMID 15363828
- [Result] O'Meara JG, Kardia SL, Armon JJ, Brown CA, Boerwinkle E, Turner ST. Ethnic and sex differences in the prevalence, treatment, and control of dyslipidemia among hypertensive adults in the GENOA study. Arch Intern Med. 2004 Jun 28;164(12):1313-8. doi: 10.1001/archinte.164.12.1313. PMID 15226165
- [Result] Turner ST, Jack CR, Fornage M, Mosley TH, Boerwinkle E, de Andrade M. Heritability of leukoaraiosis in hypertensive sibships. Hypertension. 2004 Feb;43(2):483-7. doi: 10.1161/01.HYP.0000112303.26158.92. Epub 2004 Jan 12. PMID 14718359
- [Result] Province MA, Kardia SL, Ranade K, Rao DC, Thiel BA, Cooper RS, Risch N, Turner ST, Cox DR, Hunt SC, Weder AB, Boerwinkle E; National Heart, Lung and Blood Institute Family Blood Pressure Program. A meta-analysis of genome-wide linkage scans for hypertension: the National Heart, Lung and Blood Institute Family Blood Pressure Program. Am J Hypertens. 2003 Feb;16(2):144-7. doi: 10.1016/s0895-7061(02)03248-x. PMID 12559682
- [Result] Wu X, Cooper RS, Borecki I, Hanis C, Bray M, Lewis CE, Zhu X, Kan D, Luke A, Curb D. A combined analysis of genomewide linkage scans for body mass index from the National Heart, Lung, and Blood Institute Family Blood Pressure Program. Am J Hum Genet. 2002 May;70(5):1247-56. doi: 10.1086/340362. Epub 2002 Mar 28. PMID 11923912
- [Result] Province MA, Boerwinkle E, Chakravarti A, Cooper R, Fornage M, Leppert M, Risch N, Ranade K. Lack of association of the angiotensinogen-6 polymorphism with blood pressure levels in the comprehensive NHLBI Family Blood Pressure Program. National Heart, Lung and Blood Institute. J Hypertens. 2000 Jul;18(7):867-76. doi: 10.1097/00004872-200018070-00008. PMID 10930184
- [Result] Morrison AC, Brown A, Kardia SL, Turner ST, Boerwinkle E; Genetic Epidemiology Network of Arteriopathy (GENOA) Study. Evaluating the context-dependent effect of family history of stroke in a genome scan for hypertension. Stroke. 2003 May;34(5):1170-5. doi: 10.1161/01.STR.0000068780.47411.16. Epub 2003 Apr 24. PMID 12714704